CLINICAL TRIAL: NCT00323297
Title: A Multinational, Multicentre, Randomized, Double-blind Study To Assess The Efficacy And Safety Of Oral Sildenafil 20mg Tid Or Placebo When Added To Bosentan In The Treatment Of Subjects, Aged 18 Years And Above, With Pulmonary Arterial Hypertension (Pah)
Brief Title: Assess the Efficacy and Safety of Sildenafil When Added to Bosentan in the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1481243; 2006-001464-23 (EudraCT Number); PATHWAYS (Other: Alias Study Number)
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Bosentan; Other: Placebo
- Active (Experimental)
  Interventions: Drug: Bosentan; Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Bosentan — Bosentan + Placebo for 12 weeks of the study (double blind), then 12 months open label phase (bosentan + sildenafil)
  Arms: placebo
Other: Placebo — Bosentan + Placebo for 12 weeks of the study (double blind), then 12 months open label phase (bosentan + sildenafil)
  Arms: placebo
Drug: Bosentan — Bosentan + Sildenafil for 12 weeks of the study (double blind), then 12 months open label phase
  Arms: Active
Drug: Sildenafil Citrate — Bosentan + Sildenafil for 12 weeks of the study (double blind), then 12 months open label phase
  Arms: Active

SUMMARY:
To assess the efficacy and safety of sildenafil when added to patients with PAH who are taking bosentan as all or part of their background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and over above with PAH and for which bosentan therapy is indicated according to national license
* Subjects with a mean pulmonary artery pressure of >25mmHg and a pulmonary artery wedge pressure of <15mmHg at rest via right heart catheterization within 3 years prior to randomization.
* Subjects whose baseline 6 Minute Walk Test distance is >100m and < 450m.

Exclusion Criteria:

* PAH secondary to any aetiology including congenital heart disease other than those specified in the inclusion criteria
* Subjects whose 6 Minute Walk Test may be limited by conditions other than PAH related dyspnoea or fatigue eg. claudication from vascular insufficiency or arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (6):
  - West Los Angeles VA Healthcare, Pulmonary Hypertension Program, Los Angeles, California
  - Henry Ford Hospital, Detroit, Michigan
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
- Australia (2):
  - St. Vincents Hospital, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Klinika kardiologie, Prague
- France (3):
  - Clinique des Maladies Respiratoires, Lille
  - Hopital Claude Huriez, Lille
  - Hopital Adules Brabois, Vandœuvre-lès-Nancy
- Germany (10):
  - Unfallkrankenhaus Berlin, Klinik fuer Innere Medizin, Berlin
  - II. Medizinische Klinik, Kardiologie, Angiologie und Pneumologie, Coburg
  - Universitaetsklinikum Essen, Zentrum fuer Innere Medizin, Klinik fuer Kardiologie, Essen
  - Universitaetsklinikum Giessen und Marburg GmbH, Standort Giessen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum des Saarlandes, Innere Medizin V, Homburg
  - Medizinische Klinik und Poliklinik I, Universitaetsklinikum Leipzig, Leipzig
  - Med. Klinik u. Poliklinik I der LMU Muenchen, Klinikum Grosshadern, München
  - Praxis fuer Innere Medizin, Kardiologie und Angiologie, Nuremberg
  - Missionsaerztliche Klinik Wuerzburg, Gemeinnuetzige Gesellschaft mbH, Würzburg
- Attikon Hospital, Haidari, Athens, Greece
- Israel (2):
  - Rambam Medical Center, Haifa
  - Rabin Medical Centre, Petah Tikva
- Italy (2):
  - Cardiologia, Azienda Ospedaliera Monaldi, Seconda Università di Napoli, Napoli
  - Unita' di Ipertensione Polmonare, Dipartimento di Scienze Respiratorie e Cardiovascolari, Roma
- Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan
- PVDU, Papworth Everard, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Vizza CD, Jansa P, Teal S, Dombi T, Zhou D. Sildenafil dosed concomitantly with bosentan for adult pulmonary arterial hypertension in a randomized controlled trial. BMC Cardiovasc Disord. 2017 Sep 6;17(1):239. doi: 10.1186/s12872-017-0674-3. PMID 28874133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 29 active centers in 10 countries (10 centers in Germany, 5 centers in the United States of America [USA], 3 centers in France, 2 centers in Australia, Czech Republic, Italy, and Israel, and 1 center in Greece, Taiwan and United Kingdom [UK])
Pre-assignment Details: Participants were on bosentan therapy for 3 months prior. Participants were randomized to sildenafil or placebo. Part A study was double-blind phase (12 weeks) and Part B was 12 months open-label phase. 53 and 51 participants were randomized to placebo and sildenafil arm respectively. One participant in sildenafil arm did not receive any treatment
Groups:
- Placebo: In Part A of the study: the participants received placebo three times a day (TID), in addition to their existing stable bosentan treatment (62.5 mg BID or 125 mg BID for minimum 3 months prior to randomization), for 12-Week Double-Blind Phase of the study.
  In Part B of the study: All the participants received sildenafil 20 mg TID for 12 months.
- Sildenafil: In Part A of the study: the participants received sildenafil 20 mg TID, in addition to their existing stable bosentan treatment (62.5 mg BID or 125 mg BID for minimum 3 months prior to randomization), for 12-Week Double-Blind Phase of the study.
  In Part B of the study: All the participants received sildenafil 20 mg TID for 12 months.
Period: Part A (Double Blind Randomized)
Arm/Group | Placebo | Sildenafil
Started | 53 | 50
Completed | 48 | 43
Not Completed | 5 | 7
Not completed — Reason unspecified | 0 | 1
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Unrelated adverse event | 1 | 0
Not completed — Related and Unrelated adverse event | 1 | 0
Not completed — Related adverse event | 2 | 2
Period: Part B (Open-label)
Arm/Group | Placebo | Sildenafil
Started | 48 | 43
Completed | 39 | 31
Not Completed | 9 | 12
Not completed — Death | 0 | 1
Not completed — Reason unspecified | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 3 | 1
Not completed — Adverse Event | 5 | 5
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sildenafil | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (14.14) | 55.2 (15.10) | 56.0 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 12 | 13 | 25
Six Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: Meters] — 6MWT is the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety.
  Meters | 350.38 (87.587) | 354.44 (73.121) | 352.35 (80.520)
Mean Pulmonary Artery Pressure (mPAP) [Mean (Standard Deviation); unit: Millimeter(mm) of mercury(Hg)] | 44.9 (13.33) | 46.9 (12.47) | 45.8 (12.89)
World Health Organization Functional Class in Participants with Pulmonary Arterial Hypertension [Number; unit: Participants] — Pulmonary Arterial Hypertension criteria for WHO Class: Class I (Participants with no limitation of physical activity); Class II (Participants with slight limitation of physical activity); Class III (Participants with marked limitation of physical activity); Class IV (Participants with inability to carry out any physical activity).
  Participants
    Class I | 0 | 0 | 0
    Class II | 15 | 20 | 35
    Class III | 38 | 29 | 67
    Class IV | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Distance Walked During 6 Minute Walk Time (6MWT) at Week 12
Description: 6MWT is the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) Population (Full Analysis Set) consisted of all participants who had been randomly assigned to study drug and received at least one dose of study medication. Missing values were replaced according to the last observation carried forward (LOCF) approach. Statistical analysis was carried out on LOCF values.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 53 | 50
Meters
  Change from baseline at Week 12 (n=46,44) | 17.42 (57.270) | 14.08 (63.679)
  Change from baseline at Week 12 LOCF (n=53,49) | 14.08 (57.557) | 13.62 (60.950)
Statistical Analysis 1: Comparison: Placebo vs Sildenafil; The estimated sample size was based upon the primary endpoint. A sample size of 51 subjects per treatment group was required to detect a difference of 30 meters between treatments with 80% power at a one-sided significance level of 0.05, assuming a standard deviation of 60 meters. This primary statistical analysis was carried for Week 12 data; Test type: Superiority or Other; p = 0.5802, ANCOVA — A sequential closed-testing procedure was implemented for all secondary endpoints. If no statistically significant treatment effect was found for the primary endpoint then statistical tests were not to be performed on the secondary endpoints; The mean difference in method of estimation is the difference between Sildenafil - placebo; Mean Difference (Final Values) = -2.38, 90% CI 2-sided [-21.843 to 17.087], Standard Error of Mean 11.722

2. Secondary Outcome: Number of Participants With Change From Baseline in World Health Organization (WHO) Functional Class in Participants With PAH at Week 12 LOCF
Description: WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity) to Class IV (can not perform a physical activity without any symptoms, dyspnea at rest). Improvement=reduction in functional class; deterioration = increase in functional class, no change = no change in functional class.
Time Frame: Week 12
Population: ITT Population (Full Analysis Set) consisted of all participants who had been randomly assigned to study drug and received at least one dose of study medication. Missing values were replaced according to the LOCF approach.
Measure: Number; unit: Participants
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 53 | 50
Participants
  Worsened 2 Classes | 0 | 0
  Worsened 1 Class | 1 | 0
  No Change | 45 | 39
  Improved 1 Class | 7 | 10
  Improved 2 Classes | 0 | 0
  Discontinued | 0 | 0
  Died | 0 | 1
  Missing | 0 | 0

3. Secondary Outcome: Clinical Worsening Events
Description: No survival analysis was carried out for the study due to very few events of clinical worsening. Hence, we present a summary of clinical worsening events instead.
  Events of clinical worsening were categorized as (A). Death, (B). Heart/lung transplantation, (C). Hospitalization due to pulmonary arterial hypertension (PAH), and (D). Clinical deterioration of PAH requiring additional therapy.
Time Frame: Week 12
Population: ITT Population (Full Analysis Set) consisted of all participants who had been randomly assigned to study drug and received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 53 | 50
Participants
  None | 51 | 47
  (A) | 0 | 1
  (B) | 0 | 0
  (C) | 2 | 2
  (D) | 0 | 0

4. Secondary Outcome: Change From Baseline in Borg Dyspnea Score at Week 12
Description: Borg dyspnea scale is a 10-point scale where following scores stands for severity of dyspnea: 0 (no breathlessness at all); 0.5 (very very slight [just noticeable]);
  1. (very slight);
  2. (slight breathlessness);
  3. (moderate); 4 (some what severe);
  5 (severe breathlessness); 7 (very severe breathlessness); 9 (very very severe [almost maximum]); and 10 (maximum).
Time Frame: Week 12
Population: ITT Population (Full Analysis Set) consisted of all participants who had been randomly assigned to study drug and received at least one dose of study medication. Missing values were replaced according to the last observation carried forward LOCF approach.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 53 | 50
Units on a scale
  Change from Baseline at Week 12 (n=46,43) | 0.16 (1.637) | -0.73 (1.656)
  Change from Baseline at Week 12 LOCF (n=53,49) | 0.24 (1.709) | -0.62 (1.583)

5. Secondary Outcome: One Year Survival Probability From the Start of Sildenafil Treatment.
Description: The survival probability of all participants up to 1-year post start of Sildenafil treatment; for participants who were randomized to Sildenafil, this was the week 52 from randomization, and for participants who were originally randomized to Placebo group, this was the Week 64 from Baseline (Week 52 from Week 12, when the first dose of Sildenafil was administered to these participants). Those participants who discontinued from the study prior to 1 year after start of sildenafil were considered as censored at the time of discontinuation and those who discontinued from the study post 1-year after start of sildenafil were considered as censored at the time of 1-year post start of sildenafil.
Time Frame: One year from the time of starting sildenafil
Population: ITT Population (Full Analysis Set) consisted of all participants who had been randomly assigned to study drug and received at least one dose of study medication. Missing values were replaced according to the last observation carried forward LOCF approach. The participants in placebo arm have received Sildenafil on or after Week 12.
Measure: Number (90% Confidence Interval); unit: Probability of death
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 48 | 50
Probability of death | 0.042 [0.013 to 0.127] | 0.040 [0.013 to 0.124]

6. Secondary Outcome: One Year Survival From the Start of Sildenafil Treatment.
Description: The survival status of all participants who discontinued from the study, including those participants who discontinued during the double-blind phase, was to be assessed at one year post their Week 12 visit/ End of treatment visit.
Time Frame: One year from the time of starting sildenafil
Population: as for outcome 5
Measure: Number; unit: Participants who died
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 48 | 50
Participants who died | 2 | 2

ADVERSE EVENTS:
Time Frame: From the time that the participant provides informed consent through and including 28 calendar days after the last administration of the investigational product
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Sildenafil
Serious Adverse Events (participants affected / at risk) | 23/53 | 22/50
Other Adverse Events (participants affected / at risk) | 38/53 | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | Sildenafil (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Walking distance test abnormal (Investigations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | Sildenafil (N=50)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (5)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Oedema peripheral (General disorders) | 8 (8) | 7 (7)
Bronchitis (Infections and infestations) | 5 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 7 (7)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Flushing (Vascular disorders) | 4 (4) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Palpitations (Cardiac disorders) | 3 (3) | 5 (5)
Right ventricular failure (Cardiac disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 4 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 5 (5) | 1 (1)
Weight increased (Investigations) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 3 (3)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.